CLINICAL TRIAL: NCT07358806
Title: A Phase 1 Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of OCT-598 as a Single Agent and in Combination With Standard-of-Care Treatment in Patients With Advanced Solid Tumors
Brief Title: Study to Assess the Effect of OCT-598 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oscotec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OSCO-P1401
Record Dates: First submitted 2025-12-07; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor; Breast Cancer; Head and Neck Cancer; Non-Small Cell Lung Cancer; Prostate Cancer; Gastric/Gastroesophageal Junction Cancer
Keywords: EP2/EP4 antagonist
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- PART A. OCT-598 100mg QD (Experimental): Administered orally
  Interventions: Drug: OCT-598
- PART A. OCT-598 200mg QD (Experimental): Administered orally
  Interventions: Drug: OCT-598
- PART A. OCT-598 300mg QD (Experimental): Administered orally
  Interventions: Drug: OCT-598
- PART A. OCT-598 500mg QD (Experimental): Administered orally
  Interventions: Drug: OCT-598
- PART A. OCT-598 800mg QD (Experimental): Administered orally
  Interventions: Drug: OCT-598
- PART A. OCT-598 1200mg QD (Experimental): Administered orally
  Interventions: Drug: OCT-598
- PART B. OCT-598 DL1 QD (Experimental): Administered orally, Combination with Docetaxel
  Interventions: Drug: OCT-598; Combination Product: Docetaxel
- PART B. OCT-598 DL2 QD (Experimental): Administered orally, Combination with Docetaxel
  Interventions: Drug: OCT-598; Combination Product: Docetaxel
- PART B. OCT-598 DL3 QD (Experimental): Administered orally, Combination with Docetaxel
  Interventions: Drug: OCT-598; Combination Product: Docetaxel

INTERVENTIONS:
Drug: OCT-598 — OCT-598 will be administered orally once daily.
Combination Product: Docetaxel — Docetaxel will be provided for Part B only to support the combination therapy with the standard-of-care regimen.
  Arms: PART B. OCT-598 DL1 QD; PART B. OCT-598 DL2 QD; PART B. OCT-598 DL3 QD

SUMMARY:
This is a Phase 1 study intended to determine the MTD of OCT-598 following multiple-dose therapy and to establish the RP2D for OCT-598 as a single agent, by assessing its safety and tolerability as monotherapy and in combination with standard-of-care treatments in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, ≥18 years of age (or ≥19 years according to according to the local regulatory guidance), at the time of screening
* Signed informed consent prior to any study-related procedures that are not considered standard of care
* Life expectancy >12 weeks in the opinion of the investigator
* Adequate organ and marrow function, defined as follows:

  * Absolute neutrophil count ≥1.5 × 109/L
  * Platelets ≥100,000/μL
  * Hemoglobin ≥9.0 g/dL
  * Total bilirubin <1.5 × ULN
  * ALT or AST ≤2.5 × ULN
  * Creatinine clearance calculated using the Cockcroft-Gault formula ≥60 mL/min (In equivocal cases, a 24-hour urine collection test can be used to estimate the creatinine clearance more accurately)
* LVEF >50% or within institutional values
* At least 1 measurable lesion based on RECIST version 1.1
* Cohort-specific disease requirements:

  1. Part A: patients with advanced solid tumors and no effective standard therapy option or for whom standard-of-care treatment is not available or not appropriate as per the investigator's discretion
  2. Part B: patients with advanced solid tumors who are candidates for receiving docetaxel as a single agent for their cancer treatment, including but not limited to: advanced human epidermal growth factor receptor 2-negative breast cancer, recurrent/metastatic head and neck cancer, non-small cell lung cancer, prostate cancer, or gastric/gastroesophageal cancer
* Docetaxel-appropriate (Part B): patients who have not received prior docetaxel in the advanced setting are eligible

Exclusion Criteria:

* Treatment with any IP or other anticancer therapy (including chemotherapy, antibody-drug conjugates, targeted agents, and immunotherapy) within 28 days or 5 half-lives, whichever is longer, of the first dose of study drug.
* Prior clinically significant treatment-related toxicities not resolved to Grade ≤1 or baseline (per CTCAE version 5.0) except for alopecia. Participants with stable Grade 2 peripheral neuropathy or endocrinopathies with stable endocrine replacement therapy are eligible. Patients with irreversible toxicity that is not reasonably expected to be exacerbated by study treatment (eg, vitiligo or hearing loss) may be eligible after discussion with the Sponsor.
* Prior treatment with an EP2 and/or EP4 antagonist.
* Major surgery or wide-field radiation within 28 days or limited field palliative radiation within 7 days prior to the first dose of the study drug.
* Known active central nervous system metastasis. Patients with asymptomatic previously treated brain metastasis are eligible if they are clinically stable for at least 4 weeks prior to enrollment and do not require treatment with corticosteroids.
* Treatment with systemic corticosteroids at a dose of >10 mg of prednisone or equivalent at the time of enrollment, or any other immunosuppressive medication 7 days before the first dose of the study drug. Premedication with corticosteroids prior to chemotherapy administration in the combination phase is allowed, as per the site standard of care. Systemic treatment with NSAIDs, COX2 inhibitors, or synthetic prostaglandins within 5 half-lives prior to the first dose of study drug (acetylsalicylic acid ≤160 mg/day, or 325 mg ≤3 times/week is permitted).
* Patients who are pregnant, breastfeeding, or planning to become pregnant during the study .
* Concomitant active malignancy or previous malignancy within 2 years of the time of enrollment. Patients with adequately resected basal or squamous cell carcinoma of the skin, carcinoma in situ or the cervix or breast, stage 1 prostate cancer, or other malignancy deemed to be cured by prior therapy in the judgment of the investigator may enroll regardless of the time of diagnosis.
* History of bleeding disorders, including gastrointestinal bleeding. Subjects with prior gastrointestinal bleeding due to the primary tumor, that is currently controlled, are allowed to participate.
* Mean resting corrected QT (QTc) interval using Fridericia's formula (QTcF) >470 ms, regardless of gender, or history of additional risk factors for torsades de pointes (eg, heart failure, hypokalemia, family history of long QT syndrome). Patients with left bundle block or atrial fibrillation are eligible if QTc cannot be accurately calculated provided that there is no prior history of prolonged QTc.
* For patients in Part B only: AST and/or ALT >1.5 × ULN concomitant with alkaline phosphatase >2.5 × ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability by measuring the frequency and severity of adverse events, as assessed by CTCAE v5.0 | Approximately 2 years
Incidence of Dose-Limiting Toxicities (DLTs) for Determination of the Maximum Tolerated Dose (MTD) | Approximately 2 years
Incidence of adverse events and dose-limiting toxicities used to determine the recommended Phase 2 dose (RP2D) of OCT-598 (PART B only) | Approximately 1 years

SECONDARY OUTCOMES:
To assess the maximum observed plasma concentration (Cmax) of OCT-598. | Approximately 2 years
To evaluate the effect of food on the pharmacokinetics of OCT-598 by comparing Cmax under fed and fasted conditions. | From enrollment to Cycle 1 Day -3 (PART A only)
To measure time of maximum plasma concentration (Tmax) | Approximately 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital (SNUBH), Seongnam-si
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No